CLINICAL TRIAL: NCT04421339
Title: Melatonin for Huntington's Disease (HD) Gene Carriers With HD Related Sleep Disturbance - a Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: Huntington's Disease Society of America (Other)
Responsible Party: Principal Investigator, Erin Furr Stimming, Associate Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: HSC-MS-19-1111
Record Dates: First submitted 2020-06-04; First posted 2020-06-09 (Actual); Last update posted 2023-05-15 (Actual); Status verified 2023-05

CONDITIONS: Huntington Disease
Keywords: Huntington's Disease; Melatonin
MeSH Terms: conditions — Huntington Disease | interventions — Melatonin

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Melatonin (Experimental)
  Interventions: Dietary Supplement: Melatonin
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Melatonin — Participants will receive melatonin 5 mg once a day (30 min prior to bedtime) for four weeks, followed by one-week washout before crossing-over.
  Arms: Melatonin
Other: Placebo — Participants will receive placebo once a day (30 min prior to bedtime) for four weeks, followed by one-week washout before crossing-over.
  Arms: Placebo

SUMMARY:
The purpose of the study is to evaluate the efficacy of exogenous melatonin in improving sleep quality in HD gene carriers.

ELIGIBILITY:
Inclusion Criteria:

* Verified HD mutation carriers.
* Patients who report sleep disturbance as measured by a score ≥5 on the Pittsburgh Sleep Quality Index (PSQI);
* Stable concomitant medication (no change of medication during last 30 days prior to inclusion);
* Written informed consent by prospective study participant before conduct of any trial-related procedure;
* Participant must be able to make an informed decision of whether or not to participate in the study.

Exclusion Criteria:

* Pregnant or nursing women;
* Woman of childbearing potential, not using highly effective methods of contraception such as oral, topical or injected contraception, intrauterine device (IUD), contraceptive vaginal ring, or double barrier method such as diaphragm and condom with spermicide) or not surgically sterile (via hysterectomy, ovariectomy or bilateral tubal ligation) or not at least one year post menopausal;
* Presence of any medically not controllable disease (e.g. uncontrolled arterial hypertension or diabetes mellitus);
* Use of benzodiazepines, sedating antidepressants (mirtazapine or trazodone) or sedating antipsychotics (olanzapine and quetiapine) in the previous four weeks;
* Severe cognitive disorders defined as a score < 18 on the MOCA;
* Participation in another investigative drug trial within 2 months;
* Subjects who are unlikely to be compliant and attend scheduled clinic visits as required as determined by the Investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2021-01-22 (Actual); Primary Completion 2022-09-16 (Actual); Study Completion 2022-09-16 (Actual)

PRIMARY OUTCOMES:
Change in sleep quality, as assessed by the Pittsburgh Sleep Quality Index (PSQI) | Baseline, week 5, week 9
  The PSQI is a 9-question instrument used to measure the quality and patterns of sleep in adults.
  Scoring of the answers is based on a 0 to 3 scale, whereby 3 reflects the negative extreme on the Likert Scale. A global sum of "5"or greater indicates a "poor" sleeper.

SECONDARY OUTCOMES:
Improvement in sleep quality, as assessed by the Huntington's disease (HD) sleep questionnaire | Baseline, week 5, week 9
  This questionnaire contained 45 questions that focused on different sleep-related issues such as duration, quality of sleep, abnormal nocturnal behavior and quality of life.
  The questionnaire has a total score of 19 points, scores of (0 - 3) represent the 'normal' range whilst, scores of (4 - 6) reflect 'mild' and scores of 7 and above indicate a 'significant' sleep disturbance.
Improvement in daytime somnolence, as evaluated by the Epworth Sleepiness Scale (ESS) | Baseline, week 5, week 9
  The ESS is a questionnaire designed to measure the subject's general level of daytime sleepiness.
  This scale scores from 0-24, with higher scores showing severe excessive daytime sleepiness.
Improvement in self-perceived cognitive function, as assessed by the Quality of Life in Neurological Disorders questionnaire (NeuroQOLv2.0) Cognition Function - Short Form | Baseline, week 5, week 9
  It is an 8-question instrument designed and validated to evaluate perceived difficulties in cognitive abilities (e.g., memory, attention, and decision making, or in the application of such abilities to everyday tasks (e.g., planning, organizing, calculating, remembering and learning).
  The score ranges from 0-100, with higher scores meaning a better or worse outcome according to the domain evaluated.
Improvement in global cognitive functioning, as assessed by the Montreal cognitive assessment (MoCA) | Baseline, week 5, week 9
  The MoCA was designed as a rapid screening instrument for mild cognitive dysfunction.
  Scores on the MoCA range from zero to 30, with a score of 26 and higher generally considered normal.
Improvement in quality of life, as evaluated by the Huntington's Disease Quality of Life Questionnaire (HDQoL) | Baseline, week 5, week 9
  It is a disease-specific scale containing 40 questions, with answers including different types of frequency from "never" to "all of the time".

CONTACTS AND LOCATIONS:
Overall Officials: Erin Furr Stimming, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zadegan SA, Karagas N, Tanigaki W, Duncan B, Dongarwar D, Patino J, Rocha NP, Furr Stimming E. Melatonin for Huntington's Disease (HD) gene carriers with HD-related sleep disturbance - A pilot study. Sleep Med. 2025 May;129:238-244. doi: 10.1016/j.sleep.2025.02.032. Epub 2025 Mar 4. PMID 40056659